CLINICAL TRIAL: NCT04476381
Title: Immediate Effect of Dry Needling on the Viscoelastic Properties of a Trigger Point on the Infraspinatus Muscle Measured With the MyotonPro
Brief Title: Immediate Effect of Dry Needling on Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Roch, Principal Investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MON07
Record Dates: First submitted 2020-05-27; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Shoulder Pain
Keywords: myofascial trigger points,; dry needling,; stiffness
MeSH Terms: conditions — Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: One group, one measurement of the viscoelastic properties with the MyotonPro of a single trigger point before the dry needle insertion, one measurement with the MyotonPro right after and 30 minutes later
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry needling of a trigger point in the infraspinatus muscle (Experimental): Insertion a a acupuncture type needle into a trigger point in the infraspinatus muscle on the painful side to decrease the stiffness and tone and increase the elasticity
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Insertion of a Optimed 40mm x 0.30 single use, sterile acupuncture needle into a active trigger point in the infraspinatus muscle

SUMMARY:
The immediate effects (0-30 minutes) of a dry needling intervention on a trigger point on their viscoelastic properties (tone, elasticity and stiffness)

DETAILED DESCRIPTION:
Objectives: To investigate the immediate effects of a dry needling puncture on the viscoelastic properties (tone, stiffness and elasticity) of a trigger point (TP) located in the infraspinatus muscle in participants with non-traumatic chronic shoulder pain.

Methods: Forty-eight individuals who presented non-traumatic chronic shoulder pain were recruited. The presence of a TP in the infraspinatus muscle of the painful side was confirmed by an experienced physiotherapist with a palpatory exam according to Travell and Simons criteria. The TP was marked and the viscoelastic properties including tone, stiffness and elasticity were measured with the MyotonPro device by an evaluator. After the first set of measurements (T1), an experienced physiotherapist applied a dry needling puncture to the TP with a pistoning technique to obtain a local twitch response (LTR) with an Optimed 40 x 0.30 mm single use acupuncture needle. The same set of measurements was repeated immediately after the dry needling (T2) and 30 minutes later (T3). Repeated measures ANOVA and post-hoc tests were used to assess changes in viscoelastic properties over time with a significant level set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. present with chronic shoulder pain of non-traumatic origin (rated at least 2/10 on a numeric rating scale (NRS) for more than 3 months. The pain had to be located in the shoulder area or referred in the area of the infraspinatus as described by Travell and Simons (1999);
2. have a hyperirritable spot within a palpable tight band that reproduced the participant's pain when compressed by palpation; and
3. have a body mass index (BMI) lower than 28

Exclusion Criteria:

1. diagnosis of capsulitis, cancer, or metastasis;
2. previous shoulder or thorax surgery or a mastectomy;
3. shoulder girdle bone fracture;
4. C4-C5 or C6 radiculopathy;
5. known osteoporotic profile (positive bone densitometry);
6. apparent atrophy of the infraspinatus fossa (visual interpretation) and
7. contraindications to receive a DN intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Tone in Hertz measured with a myotonometer on the trigger point | baseline
  Measurement of the tone in Hz with the myotonometer MyotonPro on the trigger point
Tone in Hertz measured with a myotonometer on the trigger point | immediately after the intervention
  Measurement of the tone in Hz with the myotonometer MyotonPro on the trigger point
Tone in Hertz measured with a myotonometer on the trigger point | 30 minutes after the intervention
  Measurement of the tone in Hz with the myotonometer MyotonPro on the trigger point
Stiffness in N/m with a myotonometer on the trigger point | baseline
  Measurement of the stiffness in N/m with the myotonometer MyotonPro on the trigger point
Stiffness in N/m with a myotonometer on the trigger point | immediately after the intervention
  Measurement of the stiffness in N/m with the myotonometer MyotonPro on the trigger point
Stiffness in N/m with a myotonometer on the trigger point | 30 minutes after the intervention
  Measurement of the stiffness in N/m with the myotonometer MyotonPro on the trigger point
Elasticity (no units: inversely proportional to the decrement of the oscillations) with a myotonometer on the trigger point | baseline
  Measurement of the elasticity with the MyotonPro
Elasticity (no units: inversely proportional to the decrement of the oscillations) with a myotonometer on the trigger point | immediately after the intervention
  Measurement of the elasticity with the MyotonPro
Elasticity (no units: inversely proportional to the decrement of the oscillations) with a myotonometer on the trigger point | 30 minutes after the intervention
  Measurement of the elasticity with the MyotonPro

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly Gaudreault, PhD, Study Director — Université de Sherbrooke
Locations (1):
- CRCHUS-Physius Lab, Sherbrooke, Quebec, Canada